CLINICAL TRIAL: NCT06279143
Title: The Diagnostic Value of Dermal Optical Coherence Tomography (D-OCT) for Clinically Suspected Basal Cell Carcinoma Lesion (BCC) in the Periocular Area
Brief Title: The Diagnostic Accuracy of Advanced Imaging in Identifying Suspected Skin Cancer (Basal Cell Carcinoma) Around the Eyes
Acronym: dOCT-pBCC
Status: Recruiting | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: dOCT-pBCC
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: BCC - Basal Cell Carcinoma; BCC; Skin Diseases; Eyelid Tumor; Eyelid Diseases
Keywords: Carcinoma, Basal Cell* / diagnostic imaging; Carcinoma, Basal Cell* / pathology; Carcinoma, Basal Cell* / surgery; Neoplasm, Glandular and epithelial; Skin neoplasm; Diagnostic imaging; Sensitivity and Specificity; Tomography, Optical Coherence* / methods; Skin Neoplasm* / surgery; Neoplasm recurrence; Eyelids / pathology; Skin diseases; Periocular; BCC
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Diseases; Eyelid Neoplasms; Eyelid Diseases; Carcinoma; Neoplasms, Glandular and Epithelial; Skin Neoplasms; Hypersensitivity; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose is to investigate the diagnostic value (sensitivity and specificity) of dermal-Optical Coherence Tomography (D-OCT, VivoSight Dx), in patients with clinically suspected BCC lesions inside the periocular region and compare these results to previous reports using D-OCT in diagnosing lesions outside the periocular area.

The Hypotheses:

* The sensitivity and specificity of D-OCT in diagnosing BCC inside the periocular region is comparable to previous reports on BCC lesions outside the periocular region when the standard D-OCT probe is used.
* The sensitivity and specificity of D-OCT in diagnosing BCC inside the periocular region is increased when the customised D-OCT probe is used.
* The sensitivity and specificity of D-OCT in diagnosing periocular BCC is comparable to punch biopsy when both standard and the customised D-OCT probes are used.
* D-OCT with the 10 and 20-millimeter standoff is capable of subtyping periocular BCC.
* The inter-observer variation in diagnosing and sub-typing periocular BCC decreases with increasing experience in the scanning procedure.
* The number of scans to correctly interpret D-OCT decreases with increasing experience in the scanning procedure.
* Delineation of periocular BCC tumour extension is possible using both D-OCT probes

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected periocular BCC.
* Biopsy-verified BCC
* Clinically suspected relapse of periocular BCC
* Age more than 18 years at baseline.
* Legally competent, able to give verbal and written consent
* Communicate in Danish verbally as well as in writing
* Willingness to participate and able to give informed consent and can comply with protocol requirements.

Exclusion Criteria:

* Anatomical circumstances that make OCT-scanning impossible, i.e., extensive scarring of eyelids, or large ulcerating crusts that hampers scanning
* Unwillingness to undergo a skin biopsy or excision of lesion.
* Inability to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive enrolment of newly referred patients under the diagnosis "clinically suspected BCC" in the periocular area
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of D-OCT in diagnosing BCC inside the periocular region, compared to previous reports on lesions outside the periocular region | March 2024-August 2026
  To assess if the sensitivity and specificity of D-OCT in diagnosing BCC inside the periocular region is comparable to previous reports on BCC lesions outside the periocular region using the standard probe

SECONDARY OUTCOMES:
Comparative diagnostic accuracy of D-OCT´s standard vs customized probe for diagnosing BCC | March 2024-August 2026
  To compare the sensitivity and specificity of each D-OCT probe for diagnosing periocular BCC, with reference to punch biopsy results.
Comparative diagnostic accuracy of D-OCT´s standard vs customized probe for subtyping BCC | March 2024-August 2026
  To compare the sensitivity and specificity of each D-OCT probe for subtyping periocular BCC, with reference to punch biopsy results.
Observer agreement in identifying presence/absence of BCC lesions, using D-OCT | March 2024-August 2026
  This measure, assesses the consistency among observers in identifying the presence or absence of BCC lesions through the utilization of D-OCT imaging.
Observer agreement in classifying BCC lesions into subtypes, using D-OCT | March 2024-August 2026
  This measure, evaluates the level of agreement among observers in categorizing BCC lesions into specific subtypes based on D-OCT imaging. Potential diagnostic features from lesion types will be tested.
Observer agreement in mapping BCC lesions prior to surgery, using D-OCT | March 2024-August 2026
  This measure, examines the agreement among observers in accurately mapping the extension of BCC lesions prior to surgery with the assistance of D-OCT imaging.
Quantification of learning curve in correctly diagnosing BCC over time with increasing experience with D-OCT | March 2024-August 2026
  This measure, quantifies the improvement in skills over time among observers in diagnosing BCC lesions using D-OCT imaging. It aims to determine the rate at which observers become adept at interpreting D-OCT images for BCC diagnosis.
Quantification of learning curve in correctly identifying BCC subtypes over time with increasing experience with D-OCT | March 2024-August 2026
  This measure, quantifies the improvement in skills over time among observers in accurately identifying different subtypes of BCC lesions using D-OCT imaging. It aims to determine the rate at which observers become adept at interpreting D-OCT images for BCC subtyping.
Quantification of skills in correctly demarcating BCC over time with increasing experience with D-OCT | March 2024-August 2026
  This measure, quantifies the improvement in skills over time among observers in precisely delineating the borders of BCC lesions prior to surgery using D-OCT imaging. It assesses the improvement in demarcation accuracy with increasing experience.
Accuracy of D-OCT in delineation of periocular BCC extension prior to surgery | March 2024-August 2026
  Evaluation af sensitivity of D-OCT imaging in delineation (mapping) of periocular BCC tumour extension - comparing findings with visible boundaries and histopathological diagnosis (considered the gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Møller, Assoc.prof., Study Director — Vejle Hospital
Locations (1):
- Department of Ophthalmology, University Hospital of Southern Denmark, Vejle Hospital, Vejle, Region of Southern Danmark, Denmark